CLINICAL TRIAL: NCT05489497
Title: Postoperative Morbidity Risk Factors After Surgical Treatment of Perforated Peptic Ulcer: a Retrospective Study of 116 Patients
Brief Title: Morbidity After Surgical Treatment of Perforated Ulcer
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Ghannouchi Mossaab, doctor, University of Monastir
Other Study IDs: perforated ulcer
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Peptic Ulcer Perforation
Keywords: Postoperative complication; Risk factor
MeSH Terms: conditions — Peptic Ulcer Perforation; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Primary closure with or without omental grafting — Primary closure with or without omental grafting

SUMMARY:
The main objective of our study is to identify the risk factors for postoperative morbidity after surgical treatment of Perforated peptic ulcer

DETAILED DESCRIPTION:
the investigators conducted a retrospective study of 116 patients, operated on for a perforated peptic ulcer, carried out in the General Surgery Department of Taher Sfar University Hospital in Mahdia over a period of 11 years 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent surgery for a perforated peptic ulcer in the General Surgery Department of Taher Sfar University Hospital in Mahdia, between January 1, 2010, and June 1, 2021, were included in this study.

Exclusion Criteria:

* patients who have medical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who presented to tahar sfar hospital for perforated ulcer
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
postoperative medical or surgical complication | baseline
  the investigators determined the number of Participants With postoperative medical or surgical complication after surgical treatement of perforated ulcer